CLINICAL TRIAL: NCT00656838
Title: Focusing Implementation to Bring Effective Reminders (FIBER)
Acronym: FIBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other); Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R01CA132709-01 (NIH); R01CA132709-01 (NIH)
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2011-10

CONDITIONS: Colorectal Cancer
Keywords: colon; rectal; cancer; screening
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Office Visits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patient has had PCP contact (letter, phone call, office visit, educational materials).
  Interventions: Behavioral: Patients receives letter, phone call, office visit, educational materials
- 2 (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Patients receives letter, phone call, office visit, educational materials — Behavioral
  Arms: 1

SUMMARY:
FIBER is 4-year study that will evaluate the implementation of a large-scale population-based colorectal cancer screening patient reminder and coordinated follow-up program. The CRC screening program began in 2007 with Kaiser Permanente Northwest (KPNW),a not-for- profit, integrated health system in Oregon and Washington. FIBER consists of 1)a practical randomized controlled trial at the start of the program, followed by 2) a longer-term cohort study as all remaining eligible patients receive the program, and 3)a qualitative evaluation. FIBER will evaluate the factors that are associated with implementation success across multiple levels: patient, primary care provider (PCP) team, specialists (gastroenterologists, general surgeons, pathologists), and other health plan staff and systems.

ELIGIBILITY:
Inclusion Criteria:

* KPNW members since 2005
* Men and women, aged 50-80 who were due for CRC screening during a 24-month period of time.

Exclusion Criteria:

* KPNW members who were part of a previous quantitative study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85289 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness and maintenance of a colon-rectal cancer screening patient reminder program.Identify patient, primary care team, and system factors important to implementation success. | Year 2, 3

SECONDARY OUTCOMES:
Create, refine, and disseminate an implementation guide for colon-rectal cancer screening reminder programs by combining the findings from the primary aim. | Years 3, 4

CONTACTS AND LOCATIONS:
Overall Officials: Adrianne C. Feldstein, MD, MS, Principal Investigator — Kaiser Foundation Hospital
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States